CLINICAL TRIAL: NCT02576730
Title: Functional Outcome Assessment After (Calcaneal) Trauma Surgey
Acronym: FACTS
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL34131.068.10/ MEC 10-3-072
Record Dates: First submitted 2015-10-05; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2010-12

CONDITIONS: Fractures; Trauma; Surgery
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fratures: patient with foot and ankle fractures and surgery with ORIF
  Interventions: Procedure: ORIF
- healthy subjects: patients without foot and ankle fracture s

INTERVENTIONS:
Procedure: ORIF — surgery for foot and ankle fractures
  Groups: Fratures

SUMMARY:
To include patient after traumatic (calcaneal) fractures for this study. They can be included to analyze gait with the OFM foot model, a non invasis model. Patient will be invited to the movement laboratory of the MUMC. Markers will be detached with dubble sided tape on anatomical points. After that gait will be recorded with infra-red camera's and an animation model will be formed. With this model further analysis can be made to range of motion between different segement of the foot. These results will be compared with patient with an arthrodesis, healthy subjects, futher questionnaires, physical examination and radiographic findings will be correlated.

DETAILED DESCRIPTION:
All subjects are asked to come to the movement laboratory of Maastricht University Medical Centre on one individual day. Before gait analyses the following characteristics were measured; height, weight, BMI, knee and ankle width (measured between the two condyles of the knee and the measured between the two malleoli of the ankle) and leg length . All measurements are performed by researchers who was trained in the examination of the foot. At least one static trial was performed with all 42 markers, with the subjects in stance phase in an anatomic neutral position. After calibrating the markers and calculating the subject-specific joint axes in the static trial, 6 markers were removed, according to the OFM protocol. After that the subjects were asked to walk barefoot in normal speed after a number of practice trials. For this speed at least 8 proper recordings were made during walking. The healthy subjects were also asked to walk in slow speed and 8 proper recordings were made during this slow-speed walking. One whole step was considered complete from heel landing (initial contact) to toe-off. A force plate was used to determine the heel-strike and toe-off phase during walking. Corrections in the axes of the knee and ankle were made if necessary and tiles were saved for further data output.

ELIGIBILITY:
Inclusion Criteria:

* patients with foot and ankle fractures

Exclusion Criteria:

* concomitant surgery for fractures of contra lateral leg/ankle or pre-existent abnormalities of the lower extremities, neurotrauma, spinal or neurological injury, pathologic fractures and people dependent in activities of daily living

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects and patients after foot and ankle trauma fracture surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Gait in Patients After foot and ankle fractures range of motion | 6 months after surgery
  To measure range of motion in the foot and ankle with the OFM (range of motion in degrees) and compare between patients with foot and ankle fractures after surgery and healthy subjects range of motion between forefoot and hindfoot, hindfoot and tibia in 3 planes representing flexion/extension, abduction/adduction, inversion/eversion

SECONDARY OUTCOMES:
To find correlations between gait, questionnaires, radiographic findings and physical examination | 6 months after surgery
  correlations between gait (OFM, see above) AOFAS score (0-100_ Foot and ankle disability index FADI 0-100 VAS pain score (0-10) Short Form 36 SF 36 physical examination range of motion in the subtalar joint (inversion/eversion) in degrees en in the ankle (flexion/extension) degrees radiographic findings (in calcaneal patients, bohlers angle, gissane's angle) in general congruency of the joint with step-off and gap